CLINICAL TRIAL: NCT07244276
Title: Comparison of Compression Continuous Suture Versus Conventional Suture for Autologous Conjunctival Implant Fixation in Primary Pterygium Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Compressed Continuous Suture and Conventional Suture in Pterygium Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: zhangyi2025
Record Dates: First submitted 2025-08-08; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Primary Pterygium
Keywords: Primary Pterygium; Compression Continuous Suture; Conventional Suture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous suture group (Other): Pterygium excision combined with autologous conjunctival transplantation was performed
  Interventions: Procedure: Compression continuous suture with suture crimping
- Intermittent suture group (Other): Pterygium excision combined with autologous conjunctival transplantation was performed
  Interventions: Procedure: Conventional Suture with suture crimping

INTERVENTIONS:
Procedure: Compression continuous suture with suture crimping — Pterygium excision combined with autologous conjunctival transplantation was performed, and the continuous suture method with pressure lines was adopted during the operation
  Arms: Continuous suture group
Procedure: Conventional Suture with suture crimping — Pterygium excision combined with autologous conjunctival transplantation was performed, and the traditional suture method was adopted during the operation
  Arms: Intermittent suture group

SUMMARY:
To compare the advantages and disadvantages of continuous suture with suture and conventional Suture in primary pterygium surgery for autologous conjunctival graft fixation

DETAILED DESCRIPTION:
Pterygium is an abnormal fibrovascular tissue hyperplasia disease that occurs in the conjunctiva. The pterygium tissue can break through the limbus of the corneosclera and grow into the cornea, causing a foreign body sensation in the eyes, astigmatism, decreased vision, and even restricted eye movement. The purpose of surgical treatment for pterygium is not only to remove the diseased tissue, but more importantly, to reduce the recurrence of pterygium after surgery. Pterygium excision combined with simple autologous conjunctival transplantation is currently the most commonly used method for treating pterygium. The recurrence rate after autologous conjunctival epithelial tissue transplantation can be reduced to 5% to 30%.

As heterogenic substances, sutures can irritate the ocular surface, aggravate postoperative inflammatory reactions and conjunctival edema or hemorrhage, delay the repair of corneal wound epithelium, lead to abnormal ocular surface function, intensify postoperative discomfort, and induce hypertrophic granuloma or cysts, etc. Moreover, these adverse reactions can also induce the recurrence of pterygium (0-26%). In addition, the longer the time interval between suture removal, The greater the difficulty of removal, the more likely some of the knots may be completely buried under the conjunctiva. Therefore, in order to alleviate the adverse reactions caused by sutures and further simplify the operation of pterygium excision surgery, many attempts have been made at home and abroad to improve and innovate the method of graft fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary pterygium according to diagnostic criteria;
2. The pterygium head invades the cornea by 2-5mm;
3. The patient agrees to the surgical treatment and signs the surgical consent form.

Exclusion Criteria:

1. History of previous eye surgery;
2. Have active ocular inflammatory lesions;
3. recurrent and pseudopterygium;
4. The patient refuses surgery or is unable to have regular follow-ups

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery | Intraoperative
  The date on which the surgery was performed
Implant stability | Postoperative follow-up was performed 1 day and 1 week after surgery
  Whether the conjunctival graft is loose or detached
Postoperative discomfort | Postoperative follow-up was performed 1 day and 1 week after surgery
  The degree of discomfort after surgery was evaluated using the VAS Pain score Scale
Stitch removal time | Postoperative follow-up was performed 1 week after surgery
  The date when the stitches were removed

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Study Director — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China